CLINICAL TRIAL: NCT03865641
Title: Effects of Virtual Reality Based Rehabilitation on Burned Hands a Prospective, Randomized, Single Blined Study
Brief Title: Effects of Virtual Reality Based Rehabilitation on Burned Hands
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hangang Sacred Heart Hospital (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HangangSHH-2
Record Dates: First submitted 2019-03-05; First posted 2019-03-07 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Hand Injuries
Keywords: burn; virtual reality
MeSH Terms: conditions — Hand Injuries; Burns

STUDY DESIGN:
Intervention Model Description: viartual reality based rehabilitation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality intervention (Experimental): Experimental group : virtual reality intervention
  Interventions: Device: Virtual reality rehabilitation
- Control group (No Intervention): conventional rehabilitation without virtual reality intervention

INTERVENTIONS:
Device: Virtual reality rehabilitation — Task-specific training has been shown to be more effective when tasks were ordered in a random practice sequence using repetition and positive feedback. VR is an interactive and enjoyable intervention. VR creates a virtual rehabilitation scene in which the intensity of practice can be systemically manipulated.
  Arms: Virtual reality intervention

SUMMARY:
Hands are the most frequent injury sites caused by burn, and appropriate rehabilitation is essential to ensure that good functional recovery is achieved. Many interventions have been developed for patients with burns; however, hand rehabilitation tools are limited. Virtual reality (VR)-based rehabilitation has proven beneficial to the functions of upper and lower extremities. To investigate VR-based rehabilitation effects on burned hands, we compare the results of VR rehabilitation group to the results of matched conventional(CON) rehabilitation group.This single-blinded, randomized, controlled trial involved 31 patients with burns and dominant right-hand function impairment. Patients were randomized into a VR or a CON group. Each intervention was applied to the affected hand for 4 weeks. Hand function was evaluated using the Jebsen-Taylor hand function test (JTT), grasp and pinch power test, and Michigan Hand Outcomes Questionnaire (MHQ). These assessments were evaluated pre-intervention and 4 weeks post-intervention.Our study results suggest that VR-based rehabilitation is likely to be as effective as conventional rehabilitation for recovering hand function in a burned hand. VR-based rehabilitation may be considered a treatment option for burned hands.

DETAILED DESCRIPTION:
Appropriate rehabilitation is important to ensure that good functional recovery is achieved. Burned hands are usually treated and managed by a multidisciplinary team at a burn center to conservatively manage hypertrophic scars. Rehabilitation of the burned hand should be initiated in the acute stages to set individualized positioning, splinting and exercise for functional activity. Frequent exercises throughout the day are more beneficial than one intensive exercise. Repeated range of motion (ROM) exercises are helpful in decreasing edema and conditioning the tissue. Despite adequate rehabilitation of the burned hand, hand functional disorders may occur. Many interventions have been developed and trialed for patients with burns; however, hand rehabilitation tools are limited and remain controversial.

Recent studies have recommended that for the functional recovery of upper extremity disorder, repetitive exercises using VR have been useful. Task-specific training has been shown to be more effective when tasks were ordered in a random practice sequence using repetition and positive feedback. VR is an interactive and enjoyable intervention. VR creates a virtual rehabilitation scene in which the intensity of practice can be systemically manipulated. This study aimed to evaluate the effects of VR-based rehabilitation on burned hands, and compare the results to those of matched CON rehabilitation in patients with burns.

ELIGIBILITY:
Inclusion Criteria:

* The patients' burn scars had re-epithelialized after aseptic care or skin graft. We included patients aged ≥18 years with a deep partial-thickness (second-degree) burn or a full thickness (third-degree) burn to their hands, with joint contracture(hand and wrist), having been transferred to the rehabilitation department after acute burn treatment, and less than 6 months since the onset of the burn injury.

Exclusion Criteria:

* patients who had fourth-degree burns(involving muscles, tendons, and bone injuries), musculoskeletal diseases(fracture, amputation, rheumatoid arthritis, and degenerative joint diseases) in the burned hand, or neurological diseases(such as peripheral nerve disorders), preexisting physical and psychologic disability (severe aphasia and cognitive impairment that could influence the intervention), and severe pain impeding hand rehabilitation.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2019-10-05 (Actual); Study Completion 2019-10-06 (Actual)

PRIMARY OUTCOMES:
hand function | 4weeks
  grip strength

SECONDARY OUTCOMES:
Michigan Hand Outcomes Questionnaire | 4weeks
  patient's perception of hand function
fine motor function | 4weeks
  Jebsen-Taylor hand function test

CONTACTS AND LOCATIONS:
Overall Officials: Cheong Hoon Seo, M.D., Study Director — Hangang Sacred Heart Hospital IRB
Locations (1):
- Hangang Sacred Heart Hospital, Seoul, Yeong-deungpo-Dong, South Korea

IPD SHARING:
Plan to Share IPD: No
after request

REFERENCES:
- [Background] Cavalcante Neto JL, Steenbergen B, Wilson P, Zamuner AR, Tudella E. Is Wii-based motor training better than task-specific matched training for children with developmental coordination disorder? A randomized controlled trial. Disabil Rehabil. 2020 Sep;42(18):2611-2620. doi: 10.1080/09638288.2019.1572794. Epub 2019 Feb 22. PMID 30794762
- [Background] Li K, Chen IM, Yeo SH, Lim CK. Development of finger-motion capturing device based on optical linear encoder. J Rehabil Res Dev. 2011;48(1):69-82. doi: 10.1682/jrrd.2010.02.0013. PMID 21328164